CLINICAL TRIAL: NCT06197113
Title: Comparison Of The Efficacies Of Intermittent Teta Burst And 10 Hz Repetitive Transcranial Magnetic Stimulation In The Treatment Of Neuropathic Pain In Patients With Spinal Cord Injury
Brief Title: Teta Burst Versus 10 Hz Repetitive Transcranial Magnetic Stimulation İn Neuropathic Pain: A Sham Controlled Comparison
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Özge Büşra Arar Batur, medical doctor, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AnkaraCHBilkent_ozgearar
Record Dates: First submitted 2023-12-26; First posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Neuropathic Pain
Keywords: Repetitive Transcranial Magnetic Stimulation; Intermittent Teta Burst Stimulation; Spinal cord injury; Depression; Pain
MeSH Terms: conditions — Neuralgia; Spinal Cord Injuries; Depression; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 10 Hz rTMS group (Active Comparator): To the patients in the high frequency (10 Hz) rTMS (n:9) group, 110% resting motor threshold (rMT), 10 Hz frequency stimulation, 5-second stimulation, and then a total of 30 trains and 1500 pulses at 25-second intervals were applied for 15 minutes while targeting the lower extremity motor area.
  Interventions: Device: Magstim Rapid2 Magnetic Stimulator
- iTBS group (Active Comparator): To the patients in iTBS group (n:9), three bursts of stimulation at 50 Hz, repeated every 200 milliseconds, were delivered for 2 seconds every 10 seconds, totaling 600 stimuli at MT intensity, applied for a duration of 200 seconds.10 sessions was applied while targeting the lower extremity motor area.
  Interventions: Device: Magstim Rapid2 Magnetic Stimulator
- Sham Group (Sham Comparator): The patients in the sham group (n:8) were given sham stimulation with a sham coil for 10 sessions.
  Interventions: Device: Magstim Rapid2 Magnetic Stimulator

INTERVENTIONS:
Device: Magstim Rapid2 Magnetic Stimulator — For TMS, the Magstim Rapid2 Magnetic Stimulator (Magstim, Whitland, Dyfed, UK) device, available in our center, was used.

SUMMARY:
Neuropathic pain is a common complication after spinal cord injury (SCI), which significantly affects the patient's quality of life and may be resistant to pharmacological treatment. In our study, we aimed to evaluate the efficacies of intermittent theta burst (iTBS) and high frequency (10 Hz) repetitive transcranial magnetic stimulation (rTMS) by comparing them with each other and with sham stimulation, in the treatment of neuropathic pain resistant to pharmacological treatment in patients with SCI.

Question 1: İs rTMS anda iTBS treatment, useful for pain severity and the effect of pain on daily functions, in the treatment of neuropathic pain in SCI Question 2: Are rTMS and iTBS treatments effective in depression in patients with neuropathic pain after spinal cord injury?

DETAILED DESCRIPTION:
Pharmacological treatments may be insufficient to limit neuropathic pain. Therefore, research continues for safe and effective new treatments. Transcranial magnetic stimulation (TMS) is a non-invasive brain stimulation method that modulates the cortical excitability of the motor area to which it is applied. Theta Burst stimulation (TBS) is a new rTMS method consisting of stimulation sequences in a special pattern. It stands out with its ability to deliver high pulses in a short time and its high capacity to induce cortical plasticity. Intermittent TBS (iTBS) and high frequency rTMS facilitate excitability in the motor area where it is applied, and this effect is used in pain treatment. Pain modulation with these methods has been tried in some studies. Therefore, repetitive magnetic stimulation of the motor cortex by these two methods may be good options for the treatment of neuropathic pain resistant to pharmacological treatment in patients with SCI.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-65,
* Traumatic/Non-traumatic spinal cord injury (>4 months),
* For >3 months, despite pharmacological treatment (no dose or medication changes have been made for at least 1 month), Brief Pain Inventory (BPI)-Part 1 average pain score is ≥4/10, neuropathic pain at the injury level and/or below (DN4 ≥4 /10) patients

Exclusion Criteria:

* Pain attributed to causes other than neuropathic pain (e.g. musculoskeletal pain, pain resulting from diabetic polyneuropathy), Having a history of epilepsy, dementia, cognitive impairment, neurodegenerative disease,
* Having a history of psychiatric illness (except reactive depression),
* Having a lesion in the brain due to vascular, traumatic, tumoral or infectious reasons,
* Having a history of alcoholism,
* Having an intracranial metallic implant,
* Having a cardiac pacemaker,
* Pregnant patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-07-11 (Actual); Study Completion 2023-07-11 (Actual)

PRIMARY OUTCOMES:
Brief Pain Inventory-Short Form (BPI-SF) | Patients were evaluated with BPI-SF before the treatment, at the end of the treatment (within the first 24 hours after the 10th session) and 4 weeks after the end of the treatment.
  Brief Pain Inventory-Short Form (BPI-SF) is designed to assess pain in sensory (pain intensity and severity) and reactive dimensions (impact on daily functioning). The BPI-SF consists of two sections. The first section evaluates the intensity of worst, least, average, and current pain using a numerical rating scale (NRS; 0-10). A response of 0 indicates no pain at all quot; and a response of 10 indicates pain as bad as you can imagine. The second section consists of seven questions that assess the impact of pain on general activity, mood, work, walking ability, sleep, relationships with others, and enjoyment of life. Responses are rated on a scale of 0 to 10. A response of 0 in the second section indicates 'does not interfere' and a response of 10 indicates 'completely interferes'. The second section total score is calculated by summing the scores of the seven questions, resulting in a score out of 70. The total score ranges from 0 to 70.

SECONDARY OUTCOMES:
Beck Depression Inventory (BDI) | Patients were evaluated with BDI before the treatment, at the end of the treatment and 4 weeks after the end of the treatment.
  The Beck Depression Inventory (BDI) is one of the most commonly used self-assessment scales to determine the level of depression. It consists of 21 items, each containing 4 options that indicate the level of the individual's mood. The patient selects the most appropriate expression for themselves. Each option is scored from 0 to 3, with 0 indicating the mildest and 3 indicating the most severe symptom. The scores from the 21 questions are added up to calculate the total score. The total score ranges from 0 to 63. It is classified as minimal (0-13), mild (14-19), moderate (20-28), and severe (29-63) depression. The Turkish validity and reliability of the scale were conducted. In this study, the BDI was used to assess the level of depression in patients with SCI.
Patient satisfaction | It was administered immediately after the end of treatment and 4 weeks after the end of treatment.
  Patient satisfaction with treatment was evaluated using a 5-point Likert scale. 1 represented 'not satisfied at all' and 5 represented very satisfied.
The level of discomfort | It was administered immediately after the end of treatment.
  4.The level of discomfort caused by the treatment was evaluated using the Visual Analog Scale (VAS). In this scale, the two ends of a 10 cm line are labeled with the extreme descriptions of the parameter to be evaluated. Although this scale is commonly used for pain assessment, it was used in our study to assess the level of discomfort. The scale ranges from 0 (no discomfort) to 10 (the most severe discomfort the patient has ever experienced in their life), and the patient is asked to mark the region that corresponds to their current condition. The distance of the marked point from the 0 point determines the patient level of discomfort.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siddall PJ. Management of neuropathic pain following spinal cord injury: now and in the future. Spinal Cord. 2009 May;47(5):352-9. doi: 10.1038/sc.2008.136. Epub 2008 Nov 11. PMID 19002150
- [Background] Lefaucheur JP, Aleman A, Baeken C, Benninger DH, Brunelin J, Di Lazzaro V, Filipovic SR, Grefkes C, Hasan A, Hummel FC, Jaaskelainen SK, Langguth B, Leocani L, Londero A, Nardone R, Nguyen JP, Nyffeler T, Oliveira-Maia AJ, Oliviero A, Padberg F, Palm U, Paulus W, Poulet E, Quartarone A, Rachid F, Rektorova I, Rossi S, Sahlsten H, Schecklmann M, Szekely D, Ziemann U. Evidence-based guidelines on the therapeutic use of repetitive transcranial magnetic stimulation (rTMS): An update (2014-2018). Clin Neurophysiol. 2020 Feb;131(2):474-528. doi: 10.1016/j.clinph.2019.11.002. Epub 2020 Jan 1. PMID 31901449
- [Background] Andre-Obadia N, Magnin M, Garcia-Larrea L. Theta-burst versus 20 Hz repetitive transcranial magnetic stimulation in neuropathic pain: A head-to-head comparison. Clin Neurophysiol. 2021 Oct;132(10):2702-2710. doi: 10.1016/j.clinph.2021.05.022. Epub 2021 Jun 20. PMID 34217600
- [Background] Cleeland CS, Ryan KM. Pain assessment: global use of the Brief Pain Inventory. Ann Acad Med Singap. 1994 Mar;23(2):129-38. PMID 8080219
- [Background] Yildirim Y, Parlar Kilic S, Eyigor S, Eyigor C, Yildirim Y, Karaman E, Oyur Celik G, Uyar M. Validity and reliability of Turkish version of the Brief Pain Inventory-Short Form for patients with chronic nonmalignant pain. Agri. 2019 Nov;31(4):195-201. doi: 10.14744/agri.2019.25901. PMID 31741339
- [Background] Richter P, Werner J, Heerlein A, Kraus A, Sauer H. On the validity of the Beck Depression Inventory. A review. Psychopathology. 1998;31(3):160-8. doi: 10.1159/000066239. PMID 9636945
- [Background] Herwig U, Satrapi P, Schonfeldt-Lecuona C. Using the international 10-20 EEG system for positioning of transcranial magnetic stimulation. Brain Topogr. 2003 Winter;16(2):95-9. doi: 10.1023/b:brat.0000006333.93597.9d. PMID 14977202
- [Background] Kobayashi M, Pascual-Leone A. Transcranial magnetic stimulation in neurology. Lancet Neurol. 2003 Mar;2(3):145-56. doi: 10.1016/s1474-4422(03)00321-1. PMID 12849236
- [Background] Huang YZ, Edwards MJ, Rounis E, Bhatia KP, Rothwell JC. Theta burst stimulation of the human motor cortex. Neuron. 2005 Jan 20;45(2):201-6. doi: 10.1016/j.neuron.2004.12.033. PMID 15664172